CLINICAL TRIAL: NCT02330497
Title: Efficacy and Safety of Radiofrequency Ablation Under Endoscopic Ultrasonography Guidance in Pancreatic Neuroendocrine and Cystic Tumor
Brief Title: Efficacy and Safety of Radiofrequency Ablation in Pancreatic Neuroendocrine and Cystic Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, MD, MSc, Société Française d'Endoscopie Digestive
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFAP
Record Dates: First submitted 2014-12-20; First posted 2015-01-05 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Tumor; Endocrine Tumor; Neoplasms, Cystic, Mucinous, and Serous
MeSH Terms: conditions — Pancreatic Neoplasms; Endocrine Gland Neoplasms; Neoplasms, Cystic, Mucinous, and Serous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency (Experimental): Procedure/Surgery Thermal Radiofrequency Ablation under endoscopic ultrasonography guidance of the pancreatic neuro endocrine tumor or mucinous cyst.
  Interventions: Procedure: Radiofrequency Ablation under EUS

INTERVENTIONS:
Procedure: Radiofrequency Ablation under EUS — Pancreatic radiofrequency ablation under endoscopic ultrasonography guidance Procedure under general anesthesia Punction of the pancreatic lesion and aspiration of the liquid if present / then thermal ablation with a 18G needle (50 W during 10 secondes) - only one session
  Other Names: Radiofrequency

SUMMARY:
Advances in conventional imaging (abdominal ultrasound, CT scan, MRI) are so great that chance to discover a incidental solid or cystic pancreatic lesion is becoming usual. Endocrine tumors have variable malignant potential depending on their size, some malignancy for lesions larger than 2 cm and indefinite for a smaller size. The branch-duct like IPMN (intraductal papillary mucinous pancreatic tumor) involving the pancreatic secondary ducts represent half of pancreatic cystic tumors and may degenerate into 5 to 10% of cases. Signs and risk of degeneration are the presence of mural nodules greater than 5 mm and size > 3 cm, although the latter criterion is discussed. Mucinous cystadenomas could degenerate between 30 and 50% of cases even though the role of size is much discussed (<4 cm). The follow-up imaging is performed using MRI and endoscopic ultrasonography (EUS). A fine needle aspiration for cytology and histology is possible and determination of biological markers is useful. But cytology is often unprofitable due to the poor cellular profile of the cystic pancreatic tumor. Once the diagnosis of suspected malignancy, the patient should be referred to the surgeon for pancreatic resection more or less extensive. But this attitude is facing a significant operative risk with up to 30% of morbidity and mortality between 1 and 3 % for cephalic resections. Some patients with high post operative risks are inoperable. For these reasons, some teams have proposed the destruction of the walls of the cyst under EUS, US or CT control by washing with absolute alcohol content of cystic tumor.

An interesting alternative endoscopic destruction would be the use of radio frequency ablation technique (RFA). RFA is a recognized technique for local tumor destruction by delivering thermal energy to obtain coagulation necrosis of the lesion. Taewong Medical ™ recently developed a radiofrequency needle EUSRA® coupled with a combo VIVA ™ generator for applying RFA sub EUS control. But no prospective study is available at this date regarding the treatment of the cystic or solid tumoral pancreatic lesion with this technique. The primary endpoint of the present study is to investigate the feasibility and safety of this guided radiofrequency probe EUS for the treatment of pancreatic endocrine tumors or inoperable pancreatic cystic tumors. The secondary objective will be the efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic neuro endocrine tumor <2 cm confirmed by pathological reading, or mucinous cystic tumor (branch duct like IPMN with nodule wall > 5 mm unresectable) or mucinous cystadenoma with unresectable wall thickening
* Unresectable patient or high operative risk
* Multidisciplinary Collaborative Meeting confirming the indication for treatment.
* Patients who consented to participate in the study
* American Society Anesthesiology classification 1, 2 or 3
* Patient affiliated to the national social security system (beneficiary or assignee)

Exclusion Criteria:

* Invasive carcinoma lesions in a patient whose clinical condition allows to consider a surgical pancreatic resection
* Severe coagulopathy (PT <50%, partial thromboplastin time > 42 sec), thrombocytopenia (<75,000 G/L), antiplatelets agent
* Patient under anticoagulant agent (NACO, heparin and warfarin)
* American Society Anesthesiology classification 4
* Patient belonging to a so-called vulnerable patient population (pregnancy, nursing, patient trust, guardianship, private patient freedom, ...)
* Women of childbearing age, including in contraception
* Pace maker
* Inability to obtain informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Safety of the pancreatic radiofrequency ablation under EUS guidance | At 3 months
  using the Cotton Classification

SECONDARY OUTCOMES:
Efficiency of the pancreatic radiofrequency ablation under EUS guidance | At month 6 and 12
  Decrease of the size of the lesion using CT-scan and tumoral response using the Response Evaluation Criteria in Solid Tumors criterion
Safety of the pancreatic radiofrequency ablation under EUS guidance | At 7 days, one month, 6 and 12 months
  using the Cotton Classification

CONTACTS AND LOCATIONS:
Overall Officials: Marc Barthet, MD, PhD, Study Chair — Assistance Publique des hôpitaux de Marseille
Locations (1):
- Barthet, Marseille, France

REFERENCES:
- [Derived] Barthet M, Giovannini M, Lesavre N, Boustiere C, Napoleon B, Koch S, Gasmi M, Vanbiervliet G, Gonzalez JM. Endoscopic ultrasound-guided radiofrequency ablation for pancreatic neuroendocrine tumors and pancreatic cystic neoplasms: a prospective multicenter study. Endoscopy. 2019 Sep;51(9):836-842. doi: 10.1055/a-0824-7067. Epub 2019 Jan 22. PMID 30669161